CLINICAL TRIAL: NCT03250559
Title: Ultrasonic Versus Fluoroscopic Guided Percutaneous Nephrolithotripsy in Pediatric Renal Stones: a Prospective Randomized Study
Brief Title: Ultrasonic vs. Fluoroscopic Guided PNL in Pediatric Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Asem Elqady, Principal investigator of urology-Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB000087618
Record Dates: First submitted 2017-07-23; First posted 2017-08-15 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pediatric Kidney Disease
Keywords: Stone disease
MeSH Terms: interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided group (Active Comparator): The group of renal stones that would have percutaneous nephrolithotomy under ultrasound guidance.
  Intervention: percutaneous nephrolithotomy.
  Interventions: Procedure: Percutaneous nephrolithotomy
- fluoroscopy guided group (Active Comparator): The group of renal stones that would have percutaneous nephrolithotomy under fluoroscopy guidance.
  Intervention: percutaneous nephrolithotomy.
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — Endoscopic kidney stone extraction technique.
  Other Names: percutaneous nephrolithotripsy (PNL)

SUMMARY:
Percutaneous Nephrolithotomy (PNL) was accepted as a treatment modality for large renal stones since 1980. Although radiation exposure during PNL is within the safe limits for expert endourologist, the mutagenic hazard is still present especially in pediatric population. Therefore, employing an alternative imaging technique during PNL would be of added advantage. So, the investigators want to compare the efficacy of ultrasound guided PNL with the conventional (fluoroscopy guided) PNL in pediatric population. If ultrasound guided PNL was as effective as conventional one, this means that many children could be protected from the variable hazards of radiation exposure.

DETAILED DESCRIPTION:
The incidence of pediatric urolithiasis varies by geographic area. Most cases of pediatric urolithiasis are associated with anatomic or metabolic abnormalities or urinary tract infection . PNL can be performed safely and effectively in children by experienced surgeons, resulting in a high stone-free rate and lower requirement for ancillary treatment. In adults, PNL is performed under fluoroscopic or ultrasound guidance. In pediatric age group, fluoroscopic guidance was preferred in most of the reported studies. However, fluoroscopy exposes the patient to radiation. The International Commission on Radiological Protection recommends that whole body exposure in adults should be limited to an effective dose of 20 mSv per year over 5 years. In young children, it is particularly important to protect the developing gonads and thyroid gland, as the long-term effects of exposing these organs to radiation are still unclear. In contrast to fluoroscopic guidance, ultrasound guidance does not expose the patient to radiation, it also can provide real-time monitoring during the puncturing procedure. The path and depth of the needle, and the anatomy in and around the kidney, are clearly visible on ultrasound examination

ELIGIBILITY:
Inclusion Criteria:

* All kidney stones in pediatric age group and indicated for PNL.

Exclusion Criteria:

* Children unfit for the procedure or non indicated for it.
* Parental refusal.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Stone free rate. | Day one post operative.
  Stone free rate (less than 4 mm residual is considered free).

SECONDARY OUTCOMES:
The need for blood transfusion. | within 24 hours of the procedure.
  Amount of transfused blood (if any) in milliliters.
Surrounding organ injury. | within first 24 hours post operative.
  Any injured surrounding organ e.g. liver, spleen or lung will be recorded with the degree of injury.
Radiation exposure. | within one hour during the procedure.
  Amount of radiation exposure (during fluoroscopy guided PNL) in millisievert (mSv).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elderwy, MD, Study Director — Assiut University
Locations (1):
- Faculty of medicine-Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng G, Zhao Z, Wan S, Zhong W, Wu W. Comparison of children versus adults undergoing mini-percutaneous nephrolithotomy: large-scale analysis of a single institution. PLoS One. 2013 Jun 24;8(6):e66850. doi: 10.1371/journal.pone.0066850. Print 2013. PMID 23826158